CLINICAL TRIAL: NCT00078923
Title: Phase II Clinical Trial of Soy Isoflavones Prior to Radical Prostatectomy
Brief Title: Soy Isoflavones in Treating Patients Who Are Undergoing Radical Prostatectomy for Stage I or Stage II Adenocarcinoma of the Prostate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDR0000353197; P30CA022453 (NIH); WSU-C-2418
Record Dates: First submitted 2004-03-08; First posted 2004-03-09 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage II prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Soybean Proteins; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Experimental): Arm I (control group): Patients receive 4 placebo capsules by mouth daily for three weeks.
  Interventions: Procedure: neoadjuvant therapy; Other: Placebo
- Soy isoflavones and placebo (Experimental): Arm II: Patients receive oral soy isoflavones (PTI G-2535) 150 mg genistein capsules + 3 placebo capsules by mouth daily for 3 weeks.
  Interventions: Dietary Supplement: soy isoflavones; Procedure: neoadjuvant therapy; Other: Placebo
- Soy Isoflavones/Placebo (Experimental): Arm III: Patients receive oral soy isoflavones (PTI G-2535) 300 mg genistein capsules + 2 placebo capsules by mouth daily for 3 weeks.
  Interventions: Dietary Supplement: soy isoflavones; Procedure: neoadjuvant therapy; Other: Placebo
- Soy Isoflavones (Experimental): Arm IV: Arm III: Patients receive oral soy isoflavones (PTI G-2535) 600 mg genistein capsules by mouth daily for 3 weeks.
  Interventions: Dietary Supplement: soy isoflavones

INTERVENTIONS:
Dietary Supplement: soy isoflavones
  Arms: Soy Isoflavones; Soy Isoflavones/Placebo; Soy isoflavones and placebo
Procedure: neoadjuvant therapy — Prostatectomy or Brachytherapy
  Arms: Placebo; Soy Isoflavones/Placebo; Soy isoflavones and placebo
Other: Placebo — Arm I: 4 placebo capsules Arm II: 3 placebo capsules Arm III: 2 placebo capsules
  Arms: Placebo; Soy Isoflavones/Placebo; Soy isoflavones and placebo

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent or delay the development of early cancer. Soy isoflavones may be effective in delaying the development of early prostate cancer.

PURPOSE: This randomized phase II trial is studying different regimens of soy isoflavones to compare how well they work in treating patients who are undergoing radical prostatectomy for stage I or stage II prostate cancer (adenocarcinoma).

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare blood/prostate biomarkers of oxidative stress and prostate cancer risk in patients with stage I or II adenocarcinoma of the prostate treated with 3 different dose levels of soy isoflavones before radical prostatectomy.
* Compare prostatic tissue biomarkers of proliferation and apoptosis in patients treated with these regimens.
* Determine the potential response, in terms of tumor and prostatic intraepithelial neoplasia grade and volume, extraprostatic extension, and serum prostate-specific antigen level, in patients treated with soy isoflavones and in those treated with placebo.
* Determine the safety of soy isoflavone supplementation in these patients.

OUTLINE: This is a randomized, double-blind, placebo-controlled, parallel-group study. Patients are stratified according to tumor stage (T1c vs T2). Patients are randomized to 1 of 4 treatment arms.

* Arm I (control group): Patients receive oral placebo once daily.
* Arm II: Patients receive oral soy isoflavones and oral placebo once daily.
* Arm III: Patients receive a higher dose of oral soy isoflavones and oral placebo once daily.
* Arm IV: Patients receive a higher dose (higher than arm III) of oral soy isoflavones once daily.

In all arms, treatment continues for 2-6 weeks (depending on the time from study entry to planned surgery) in the absence of unacceptable toxicity. All patients then undergo radical prostatectomy.

Patients are followed at 1 week.

PROJECTED ACCRUAL: A total of 100 patients (25 per treatment arm) will be accrued for this study within 12.5 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the prostate

  * Stage T1c or T2
  * Disease confined to the prostate gland
* Planning to undergo radical prostatectomy within the next 3-4 weeks

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* ALT and AST less than 2 times upper limit of normal (ULN)
* Alkaline phosphatase less than 2 times ULN

Renal

* Not specified

Other

* Fertile patients must use effective barrier contraception
* Medically cleared for surgery
* No concurrent thyroid disease

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior biological therapy for prostate cancer
* No concurrent biological agents

Chemotherapy

* No prior chemotherapy for prostate cancer
* No concurrent chemotherapy

Endocrine therapy

* No prior hormonal therapy for prostate cancer
* No concurrent thyroid hormone replacement medication
* No concurrent hormonal therapy

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* At least 3 months since prior high-dose nutritional supplements
* No concurrent regular use (more than once weekly) of soy products greater than 50 g of soy protein or 50 mg of soy isoflavone
* No concurrent high-dose nutritional supplements

  * Standard-dose single multivitamin tablet (e.g., Centrum™) allowed
* No concurrent herbs
* No concurrent soy foods
* No other concurrent isoflavone supplements
* No other concurrent antineoplastic agents

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2001-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Oxidative DNA damage as measured by 5-hydroxymethyluridine level | at 3 weeks
Lipid oxidation as measured by 8-isoprostane level | at 3 weeks

SECONDARY OUTCOMES:
Tumor size, grade, and extension | at 3 weeks
Prostate-specific antigen and prostatic intraepithelial neoplasia grade | at 3 weeks
Biomarkers of cell growth, differentiation, and apoptosis | at 3 weeks
Toxicity as measured by number and grade of adverse events | at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Omer Kucuk, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States